CLINICAL TRIAL: NCT06821763
Title: Effect of Calcium Hydroxide on Post Operative Pain Severity in Single Rooted Teeth with Symptomatic Apical Periodontitis
Brief Title: To Measure Post Operative Pain Severity by Using Two Different Intra Canal Medicaments Calcium Hydroxide and Triple Antibiotic Paste in Teeth with Single Roots and Periapical Disease Called Apical Periodontitis
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Komal Ashraf Khan (Other)
Responsible Party: Sponsor-Investigator, Komal Ashraf Khan, Post Graduate Trainee, Margalla Institute of Health Sciences
Organization: Margalla Institute of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DK/248/24
Record Dates: First submitted 2025-01-20; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-09

CONDITIONS: Apical Periodontitis; Irreversible Pulpitis with Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A( calcium hydroxide) (Active Comparator): patients receiving calcium hydroxide as intra canal medicament
  Interventions: Drug: Calcium Hydroxide Intracanal medication
- Group B( Triple Antibiotic Paste) (Active Comparator): Patients receiving triple antibiotic paste as intra canal medicament
  Interventions: Drug: triple antibiotic paste (TAP)

INTERVENTIONS:
Drug: Calcium Hydroxide Intracanal medication — non setting calcium hydroxide(CH) mixed with normal saline and placed as intra canal medicament during first visit of root canal treatment. effectiveness measured after 48hrs, 72hrs and 96hrs
  Arms: Group A( calcium hydroxide)
Drug: triple antibiotic paste (TAP) — mix metronidazole, ciprofloxacin and minocycline in ratio 1:1:1 with normal saline and placed as intra canal medicament during first visit of root canal treatment.
  Arms: Group B( Triple Antibiotic Paste)

SUMMARY:
* The aim of this study is to compare post operative pain effectiveness between two most commonly available intra canal medicaments that are Triple Antibiotic Paste and Calcium Hydroxide during root canal treatment of single rooted teeth with symptomatic apical periodontitis.
* Patients visiting OPD will be selected after fulfilment of inclusion criteria and randomly divided into two groups i.e group A patients receiving calcium hydroxide and group B with patients receiving Triple Antibiotic Paste as intra canal medicaments
* Patient will be called at 48hrs 72hrs and 96hrs postoperatively.
* Effectiveness of intra canal medicaments will be measured as no mild moderate severe on visual analogue scale(VAS).

DETAILED DESCRIPTION:
* This randomized control study is done to compare post operative pain effectiveness of two medicaments that are triple antibiotic paste (TAP)(ciprofloxacin, metronidazole and minocycline in ratio 1:1:1) and calcium hydroxide(CH) during root canal treatment of single rooted teeth with symptomatic apical periodontitis.
* Calcium hydroxide being strong base exerts antimicrobial efficiency in reducing and eliminating microorganisms in entire root canal system
* TAP is efficient against calcium hydroxide resistant bacteria called as enterococcus faecalis and provides antimicrobial efficiency to inner depths of root canal up to 400 microns.
* This study will add further to literature regarding better intracanal medicament among two most widely used.
* Sample size includes total 180 participants having two groups each containing 90.
* Inclusion criteria have patients with age group 12-45, single rooted teeth, having symptomatic apical periodontitis, patients fulfilling international associates definition of pain
* Exclusion criteria includes patients having allergies, unable to take medications, medical conditions like diabetes etc, pregnant patients, teeth with tooth abnormalities like dilacerations open apices etc
* Patients will be selected from OPD after fulfilment of inclusion criteria randomly divided into two groups using lottery method
* Group A receiving calcium hydroxide group B receiving triple antibiotic paste
* Patients will be called post operatively after 48hrs 72hrs and 96hrs
* Post operative pain effectiveness will be measured as no mild moderate and severe on visual analogue scale (VAS)
* The data will be analyzed in statistical software SPSS v 25. Chi square test will be applied to compare effectiveness in both groups keeping p value less than 0.05 as significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders having age 12-45 years
* Newly diagnosed cases fulfilling the criteria of INTERNATIONAL ASSOCIATES FOR THE STUDY OF PAIN definition of pain.
* A Single rooted teeth (Anterior or Posterior)
* Teeth with symptomatic apical periodontitis
* Teeth with necrotic pulp that gave a negative response to vitality testing.

Exclusion Criteria:

* Patients who have allergies, sensitivity or unable to take medications, periodontal disease, acute endodontic or periodontal abscess, requiring prophylactic antibiotics, systemic diseases like hypertension, diabetes, liver dysfunction renal failure and mental disabilities were excluded.
* Pregnant ladies or patients on nursing were also excluded from the sample.
* Teeth with anatomical difficulties such as open apices.
* Teeth with severe dilacerations, calcified canals, occlusal interferences, chronic periodontitis, internal/external root resorption.
* Patients with serious medical illness, systemic disorders, immunocompromised diseases such as AIDS or HBV.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
post operative pain | 6 months
  post operative pain measured through visual analogue scale( VAS) from readings no pain 0, mild taken as 0-2, moderate as 2-5, severe taken as 5-10

CONTACTS AND LOCATIONS:
Locations (1):
- Margalla Institute Of Health Sciences Quaid e Azam Avenue, Gulraiz phase 3, Gulraiz housing scheme Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No